CLINICAL TRIAL: NCT05904236
Title: Phase 1 First-in-Human Dose Escalation and Expansion Study to Assess Safety and Tolerability of Intravenous Administration of ICVB-1042 in Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability of Intravenous Administration of ICVB-1042
Acronym: ICVB-1042
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Demonstrated Clinical Activity
Sponsor: IconOVir Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-CLN01
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Patients With Advanced Solid Tumors
Keywords: Oncolytic virus; First in human; Relapsed solid tumor; Refractory solid tumor; Tumor biopsy; Novel therapy; Metastatic; Previously treated
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Escalating doses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICVB-1042 (Experimental): Part A: Dose escalation Part B: Dose expansion
  Interventions: Drug: Treatment with ICVB-1042 administered intravenously

INTERVENTIONS:
Drug: Treatment with ICVB-1042 administered intravenously — Part A Dose Escalation to assess safety and tolerability of ascending dose levels, define the maximum tolerated dose (MTD), and expansion dose(s) Part B Dose Expansion to further assess safety and tolerability of 1 or more dose levels

SUMMARY:
Study to evaluate the safety and tolerability of intravenous ICVB-1042

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with relapsed or refractory locally advanced or metastatic solid tumors who have progressed on or after at least one prior line of standard of care therapy including immune checkpoint inhibitors and targeted therapies for known molecular alterations if present
* Measurable disease according to RECIST v1.1
* ECOG Performance Status 0 or 1
* Life expectancy of at least 3 months

Exclusion Criteria:

* Prior SOC or other treatment with a biologic (eg, mAb) within 28 days prior to dosing or 5×half-life, whichever is longer from investigational therapy
* Major surgical procedures within 28 days prior to dosing
* Limited field irradiation for palliation within 14 days prior to dosing
* Anti-viral agents, vaccinations within 28 days prior to dosing
* Known central nervous system (CNS) metastases unless adequately treated and clinically stable without steroids for ≥14 days
* Leptomeningeal carcinomatosis
* Pulmonary lymphangitic spread of cancer
* History of clinically significant cardiovascular abnormalities
* Known active infection requiring systemic antibiotic therapy or systemic antifungal therapy
* Known active HIV, hepatitis B or C, or other active viral disease
* Known hematologic malignancies (requiring or not requiring active therapy).
* Requirement for immunosuppressive therapy (ie, prednisone equivalent of >10 mg/day)
* Women who are pregnant or lactating
* Oxygen saturation measured with Pulse oximeter <90% and/or on supplemental O2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Safety of intravenous ICVB-1042 | From dose administration through 12 weeks
  Assessment of treatment-emergent dose limiting toxicity

SECONDARY OUTCOMES:
Concentration profile of ICVB-1042 in plasma | Up to 48 hours after drug infusion
Determine immunogenicity of ICVB-1042 | From dose administration through 12 weeks
  Assessment of anti-drug antibody titer

OTHER OUTCOMES:
Evaluate shedding of ICVB-1042 | At study visits from dose administration through 12 weeks
  ICVB-1042 concentration in urine, feces, and saliva
Tumor response by RECIST criteria | Day 57
  Number of patients with complete response, partial response, stable disease or progressive disease will be assessed by tumor imaging
Concentration of ICVB-1042 in tumor biopsy | Day 57
  Measurement of ICVB-1042 in biopsy samples
Number of patients with immunoreactivity to ICVB-1042 administration | At study visits from dose administration through 12 weeks
  Evaluation of cytokine changes from baseline
Number of patients with changes in cell-free tumor DNA | At study visits on Day 1, Day 10, Day 29, Day 57, Day 85 or Early Termination visit
  Assessment of tumor DNA in plasma
Evaluate viral replication | At study visits from dose administration through 12 weeks
  Levels of viral proteins in plasma
Viral titer of ICVB-1042 | At study visits from dose administration through 12 weeks
  Evaluation of infectivity from plasma and saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Julie Maltzman, MD, Study Director — IconOVir Bio
Locations (10):
- United States (10):
  - California Cancer Associates, San Marcos, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - NYU Langone Health, Perlmutter Cancer Center, New York, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolina BioOncology, Huntersville, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Next Oncology, Dallas, Irving, Texas
  - Next Oncology, San Antonio, San Antonio, Texas
  - Next Oncology, Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kato Y, Rice N, Pokrass M, Jeong J, Rodriguez R, Field JJ, Nowyhed H. Nonclinical characterization of ICVB-1042 as a selective oncolytic adenovirus for solid tumor treatment. Commun Biol. 2024 Sep 13;7(1):1132. doi: 10.1038/s42003-024-06839-6. PMID 39271928